CLINICAL TRIAL: NCT06065176
Title: Booster Epidemiological Evaluation of Health, Illness and Vaccine Efficacy Study: Randomized Trial to Compare the Clinical Efficacy of Novavax vs. mRNA COVID-19 2023-2024 Updated Vaccines Among Adults in the United States
Brief Title: The Efficacy of the 2023-2024 Updated COVID-19 Vaccines Against COVID-19 Infection
Acronym: BEEHIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarang K. Yoon, DO, MOH (Other)
Collaborators: Westat (Other); Novavax (Industry)
Responsible Party: Sponsor-Investigator, Sarang K. Yoon, DO, MOH, Associate Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00172738
Record Dates: First submitted 2023-09-29; First posted 2023-10-03 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: COVID-19; Vaccine-Preventable Diseases; SARS CoV 2 Infection; Upper Respiratory Tract Infection; Upper Respiratory Disease
Keywords: COVID-19 vaccines; Rapid antigen test; SARS-CoV-2; Vaccine Efficacy; Real World Evidence
MeSH Terms: conditions — COVID-19; Vaccine-Preventable Diseases; Respiratory Tract Infections; Respiration Disorders | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Intervention Model Description: This randomized, three arm, active comparator trial will compare the clinical efficacy of a single dose of the Novavax 2023-2024 updated COVID-19 vaccine (Arm 1) with a single dose of the Pfizer mRNA 2023-2024 updated COVID-19 vaccine (Arm 2) as well as non-vaccinated comparison group (Arm 3). The participants who elect to receive a 2023-2024 updated COVID-19 vaccine are randomized into the Novavax (Arm 1) or Pfizer mRNA (Arm 2) vaccine groups. The non-vaccinated comparison group is nonrandomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will elect whether they are in the vaccinated group or decline to be in the vaccinated group. So, all participants will be aware of their group assignment. However, those participants in the vaccinated group as well as study investigators will be blinded to study arm assignments within the vaccinated group. A limited number of study staff handling and administering the vaccines will be aware of vaccine assignment and will be trained not to divulge vaccine assignment information to the investigator and study team. Study staff administering vaccine will not be involved with study surveillance to avoid involvement with measurement of study outcomes. The study will provide electronic documentation confirming that participants received one of the study vaccines (without indicating which vaccine) with date of vaccine administration. The electronic documentation of vaccine administration will be password protected to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Novavax COVID-19 booster (Active Comparator): Participants will receive a single dose (0.5 ml) of study vaccine Novavax COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
  Interventions: Biological: Novavax COVID-19 vaccine (2023-2024 formula XBB containing)
- Pfizer COVID-19 booster (Active Comparator): Participants will receive a single dose (0.3 ml) of study vaccine Pfizer mRNA COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
  Interventions: Biological: Pfizer COVID-19 mRNA vaccine (2023-2024 formula XBB containing)
- Non-boosted comparison group (No Intervention): Participants will not receive a dose of the study vaccine.

INTERVENTIONS:
Biological: Novavax COVID-19 vaccine (2023-2024 formula XBB containing) — Participants will receive a single dose of the Novavax vaccine.
  Arms: Novavax COVID-19 booster
Biological: Pfizer COVID-19 mRNA vaccine (2023-2024 formula XBB containing) — Participants will receive a single dose of the Pfizer vaccine.
  Arms: Pfizer COVID-19 booster

SUMMARY:
The purpose of this research study is to find out how well two different 2023-2024 updated COVID-19 vaccines protect people from COVID-19 (the disease caused by the SARS-CoV-2 virus), and to determine if getting a 2023-2024 updated vaccine provides better protection from COVID-19 than not getting a vaccine.

If the participant chooses to get a 2023-2024 updated COVID-19 vaccine as part of this study, they will have a 50/50 chance of receiving either the Novavax or Pfizer mRNA vaccine.

If the participant decides not to get a 2023-2024 updated COVID-19 vaccine, the participant can still participate in other study activities.

STUDY ACTIVITIES:

* An online enrollment survey
* An in-person enrollment visit
* Weekly online surveys for 20 weeks
* Weekly COVID-19 tests for 20 weeks
* Additional online surveys if you have COVID-19 symptoms or tested positive for COVID-19.
* Additional COVID-19 tests if you have COVID-19 symptoms or tested positive.
* Online survey questions in the middle and at the end of the study

DETAILED DESCRIPTION:
For the BEEHIVE Study, UT seeks to enroll 1,500 participants living in the greater Salt Lake City area during the upcoming 2023-2024 COVID-19 season. Participants who intend to get vaccinated with the 2023-2024 updated COVID-19 vaccine (n=1200) will be randomized into the NVX vaccine group or the Pfizer mRNA vaccine group. Participants will be randomized 1:1 to receive 1 dose of the NVX vaccine versus 1 dose of the Pfizer mRNA vaccine from October to December 2023 (dates may vary slightly based on vaccine availability). Participants who decide not to receive a 2023-2024 updated COVID-19 vaccine during this period will be placed in a non-randomized comparison group (n=300).

Participants in all three study arms will complete an online enrollment survey and will self-schedule an in-person enrollment visit. During the visit, all participants will receive a supply of at-home rapid antigen tests for SARS-CoV-2 infection. Those who choose to be in the vaccinated group will also receive either the Novavax vaccine or the Pfizer mRNA vaccine at random. On the first, second, and seventh day after receiving the vaccine, participants will complete an online post-vaccination survey. Beginning after the enrollment visit for a period of 24 weeks, all participants will complete a weekly rapid at-home test and a weekly online survey that surveils for COVID-like illness (CLI)-associated SARS-CoV-2 virus infection, defined as symptoms in the past 7 days including: fever; chills; malaise; fatigue; headache; cough; shortness of breath; sore throat; runny nose or nasal congestion; nausea or vomiting; diarrhea; muscle or body aches; or change in smell or taste. Participants will upload a photo of each weekly test result to the study portal. Those who report new CLI symptoms and those who test positive on their at-home test will complete additional online surveys concerning their illness, as well as another at-home test on the first and third day after the original test. Additionally, all participants will complete a mid- and end-of study survey about their work, health, and opinions about COVID-19, and any COVID-19 and influenza vaccines received. Finally, participants who tested positive for COVID-19 during the study or who had COVID-19 symptoms but did not test positive will complete an online survey about the duration of symptoms and impact on their health. By Summer 2024, study staff will inform participants when the weekly surveys will end and when to stop testing. At the end of the study, participants in the vaccinated group will be notified of which study vaccine they received.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Previously received ≥ 2-doses of US FDA-authorized mRNA vaccines
* Comfortable reading and responding to text messages and emails sent in English or having an interpreter assist them
* Plan to remain in the greater Salt Lake City area for the next 12 months
* Daily access to the internet (via cell phone, laptop, desktop, or tablet) and a phone with text messaging capabilities
* Willingness to complete weekly symptom and illness surveillance surveys sent via text and email
* Willingness to complete an online survey at enrollment, mid-study, and end-of-study surveys
* Willingness to be contacted periodically by study staff via text, email, and/or telephone as part of study activities
* Willingness to self-collect rapid antigen tests (RAT; approved by FDA EUA for COVID-19 detection) weekly and when prompted for study purposes, and to send results via the study portal
* Willingness to self-collect additional rapid antigen test (approved by FDA EUA for COVID-19 detection) if experiencing a qualifying symptomatic illness or upon RAT-confirmation of an asymptomatic infection
* Willingness to attend in-person visit to receive supply of rapid antigen tests and training on their use (all participants) and to receive a COVID-19 booster (if in randomized group)

Exclusion Criteria:

* Lives with another person who is already enrolled in this study as reported by the subject on the Eligibility Survey (Appendix C. Eligibility Survey)
* Previous hypersensitivity reaction to the study vaccines as reported by the subject on the Eligibility Survey (Appendix C. Eligibility Survey)
* Recent infection [Real time Reverse Transcription Polymerase Chain Reaction assay (RT-PCR) and/or RAT confirmed infection ≤ 90 days of trial vaccine administration
* Receipt of a COVID-19 vaccine within ≤ 90 days of trial vaccine administration
* Participation in other vaccine trials
* Medical history of immunosuppression
* Receipt of J&J vaccine prior to study enrollment
* Receipt of any investigational prevention therapies for SARS-CoV-2 infections, such as prophylactic antiviral medications or other immune system modifying interventions within ≤ 90 days of trial vaccine administration
* Unwillingness to provide electronic consent
* Unwillingness to self-report occupation, work responsibilities, and prior COVID-19 illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1188 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarang K Yoon, DO, Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon SK, Ellsworth GL, Battan-Wraith S, Phillips AL, Fink RV, Griffin J, Rowley EAK, McKell J, Smith AS, Campbell R, Williams J, Ball SW, Zhao H, Warren B, Rousculp MD, Thiese MS. Real-World Effectiveness and Noninferiority Evaluation and Comparison of Messenger RNA-Based and Protein-Based COVID-19 Vaccines: Protocol for the BEEHIVE Randomized Study With a Hybrid Effectiveness Design. JMIR Res Protoc. 2026 Jan 27;15:e80858. doi: 10.2196/80858. PMID 41592795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The BEEHIVE trial enrolled and monitored participants from 22 November 2023 through 9 September 2024. 5590 participants were screened.
Pre-assignment Details: 1188 total participants enrolled.
Groups:
- Novavax COVID-19 Booster: 452 participants received a single dose (0.5 ml) of study vaccine Novavax COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
- Pfizer COVID-19 Booster: 457 participants received a single dose (0.3 ml) of study vaccine Pfizer mRNA COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
- Non-boosted Comparison Group: 279 participants did not receive a dose of the study vaccine.
Period: Overall Study
Arm/Group | Novavax COVID-19 Booster | Pfizer COVID-19 Booster | Non-boosted Comparison Group
Started | 452 | 457 | 279
Completed | 437 | 440 | 266
Not Completed | 15 | 17 | 13
Not completed — Lost to Follow-up | 11 | 11 | 10
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — No longer met eligibility requirements to continue participation. | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novavax COVID-19 Booster | Pfizer COVID-19 Booster | Non-boosted Comparison Group | Total
Number analyzed (Participants) | 452 | 457 | 279 | 1188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 2 | 10
  Between 18 and 65 years | 409 | 406 | 246 | 1061
  >=65 years | 40 | 46 | 31 | 117
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex Assigned at Birth: Female | 248 | 250 | 147 | 645
  Sex Assigned at Birth: Male | 203 | 206 | 132 | 541
  Sex Assigned at Birth: Prefer Not to Answer | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 1 | 7
  Asian | 13 | 23 | 15 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 7 | 5 | 1 | 13
  White | 393 | 394 | 241 | 1028
  More than one race | 34 | 25 | 16 | 75
  Unknown or Not Reported | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 49 | 25 | 128
  Not Hispanic or Latino | 398 | 408 | 254 | 1060
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic SARS-CoV-2 Infections Between Randomized, Study-vaccinated Participants and the Comparator Group
Description: Difference in the number of symptomatic SARS-CoV-2 infections between randomized, study-vaccinated participants and the comparator group who did not receive an updated COVID-19 vaccine (2023-2024 formula).
Time Frame: 24 weeks after enrollment
Population: mITT population. Combining both vaccinated arms in a single group most appropriately represents the study's primary objective. The two vaccinated arms are assessed relative to each other in the study's secondary objective.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Booster Comparator Group: 279 participants who consented to enrollment but declined receipt of a study vaccine dose.
- Randomized Group: 909 were randomized into the protein subunit (N=452) and mRNA (N=457) groups.
  Randomized participants received a single intramuscular dose of either study vaccine (0.3 mL for mRNA and 0.5 mL for protein subunit) in the deltoid.
Arm/Group | Non-Booster Comparator Group | Randomized Group
Number analyzed (Participants) | 278 | 898
Participants | 48 | 94

2. Secondary Outcome: Number of Symptomatic SARS-CoV-2 Infections Between the Protein Subunit and mRNA Vaccine Groups.
Description: Difference in the number of symptomatic SARS-CoV-2 infections between the protein subunit and mRNA vaccine groups.
Time Frame: 24 weeks after study enrollment
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- Protein Subunit: Participants received a single dose (0.5 ml) of study vaccine Novavax COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
- mRNA: Participants will receive a single dose (0.3 ml) of study vaccine Pfizer mRNA COVID-19 vaccine, 2023-2024 formula (XBB containing) in the deltoid muscle of the arm.
Arm/Group | Protein Subunit | mRNA
Number analyzed (Participants) | 444 | 454
Participants | 52 | 42

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 24 weeks
Arm/Group | Novavax COVID-19 Booster | Pfizer COVID-19 Booster | Non-boosted Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/452 | 0/457 | 0/279
Serious Adverse Events (participants affected / at risk) | 1/452 | 5/457 | 0/279
Other Adverse Events (participants affected / at risk) | 401/452 | 436/457 | 0/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novavax COVID-19 Booster (N=452) | Pfizer COVID-19 Booster (N=457) | Non-boosted Comparison Group (N=279)
Infections due to complications of surgery (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) — Participants self-reported hospitalization due to infections that occurred secondary to infections unrelated to study participation.
Serious injuries due to auto accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Participant self-reported several severe injuries requiring prolonged hospitalization as a result of an auto accident.
Hospitalization due to mental health crisis (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) — Participant self-reported hospitalizations due to mental health
Emergency Cesarean Section due to premature labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) — Participants reported requiring emergency C-section due to premature labor during study participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novavax COVID-19 Booster (N=452) | Pfizer COVID-19 Booster (N=457) | Non-boosted Comparison Group (N=279)
Injection Site Pain (Musculoskeletal and connective tissue disorders) | 277 (277) | 382 (382) | 0 (0)
Injection Site Swelling (Musculoskeletal and connective tissue disorders) | 51 (51) | 113 (113) | 0 (0)
Injection Site Tenderness (Musculoskeletal and connective tissue disorders) | 337 (337) | 405 (405) | 0 (0)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 146 (146) | 240 (240) | 0 (0)
Fatigue (Immune system disorders) | 175 (175) | 251 (251) | 0 (0)
Fever (Immune system disorders) | 13 (13) | 40 (40) | 0 (0)
Joint Pain (Immune system disorders) | 48 (48) | 95 (95) | 0 (0)
Malaise (Immune system disorders) | 84 (84) | 177 (177) | 0 (0)
Nausea (Immune system disorders) | 26 (35) | 42 (55) | 0 (0)
Headache (Immune system disorders) | 121 (121) | 168 (168) | 0 (0)

LIMITATIONS AND CAVEATS:
These results are preliminary; analyses are ongoing, and the findings have not yet been published.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT06065176/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT06065176/SAP_001.pdf